CLINICAL TRIAL: NCT06858306
Title: SPHERE Per-AF Post-Approval Study, an Addendum to the Affera Global Registry
Brief Title: SPHERE Per-AF Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: SPHERE Per-AF PAS
Record Dates: First submitted 2025-02-26; First posted 2025-03-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Persistent Atrial Fibrillation
  Interventions: Device: Sphere-9™ Catheter and Affera™ Ablation System

INTERVENTIONS:
Device: Sphere-9™ Catheter and Affera™ Ablation System — De novo pulmonary vein isolation procedure using commercially available Sphere-9™ Catheter and Affera™ Ablation System

SUMMARY:
SPHERE Per-AF Post-Approval Study is a prospective, multi-center, non-randomized, observational trial. Subjects will be treated with the Sphere-9™ Catheter and Affera™ Ablation System and followed through 36 months.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the long-term effectiveness and safety of the Sphere-9™ Catheter and Affera™ Ablation System in a post-approval setting for the treatment of drug refractory, recurrent, symptomatic, persistent AF (episode duration less than one year).

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of recurrent symptomatic persistent AF (continuous AF sustained longer than 7 days but less than 12 months)
2. Refractory (i.e. not effective, not tolerated, or not desired) to at least one Class I or III antiarrhythmic drug (AAD)
3. Patient is ≥ 18 years of age
4. Planned de novo pulmonary vein isolation procedure using commercially available Sphere-9™ Catheter and Affera Ablation System
5. Patient is willing and able to comply with study requirements and give informed consent

Exclusion Criteria:

1. Long-standing persistent AF (continuous AF sustained >12 months)
2. Prior left atrial catheter or surgical ablation
3. Life expectancy <36 months
4. Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
5. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study not pre-approved by Medtronic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older with a planned de novo procedure using commercially available Sphere-9™ Catheter and Affera™ Ablation System.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Objective | Through 180 days Post-Procedure
  Estimate the primary safety adverse event (AE) rate for ablation using the Sphere-9™ Catheter and Affera™ Ablation System.
Primary Effectiveness Objective | Through 36 months Post-Procedure
  Estimate the 36-month freedom from atrial fibrillation (AF), atrial tachycardia (AT) or atrial flutter (AFL) recurrence following ablation procedure using the Sphere-9™ Catheter and Affera™ Ablation System.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, New York, New York
  - OhioHealth, Columbus, Ohio
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Texas Health Resources, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Centra Medical Group Stroobants Cardiovascular Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No